CLINICAL TRIAL: NCT05804435
Title: Prospective Multi-center Study Using a Bronchoscopic Ultrasound-Guided Needle Biopsy System With Real-time Visualization in Endobronchial Lesions, Peripheral Lung Nodules, or Lung Masses
Brief Title: iNod™ Ultrasound-Guided Needle Biopsy System Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: E7186
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Solitary Pulmonary Nodule; Multiple Pulmonary Nodules; Biopsy, Fine-Needle
Keywords: Post-Market; Pulmonary Lesions; iNod; R-EBUS
MeSH Terms: conditions — Solitary Pulmonary Nodule; Multiple Pulmonary Nodules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- iNod™ System (Experimental): Subjects with a qualifying lung lesion will have a standard of care Transbronchial Needle Aspiration using the the iNod™ System
  Interventions: Device: iNod™ System

INTERVENTIONS:
Device: iNod™ System — The iNod™ Ultrasound Imaging System enables visualization of endobronchial lesions, peripheral lung nodules, or lung masses (referred to as lesions) using R-EBUS and performance of lung biopsy under direct R-EBUS visualization.
  Other Names: iNod™ Ultrasound Imaging System; iNod™ SUD

SUMMARY:
The purpose of this study is to collect information on the iNod™ System's safety and ability to see the iNod™ biopsy needle in real-time in endobronchial lesions, peripheral lung nodules, or lung masses.

DETAILED DESCRIPTION:
This post-market study intends to further demonstrate the ability and safety of the iNod™ Ultrasound Guidance System and iNod™ Ultrasound Biopsy needle to perform transbronchial needle biopsy of endobronchial lesions, peripheral lung nodules, or lung masses under real-time ultrasound visualization. This is a prospective, multi-center case series of standard of care peripheral lung nodule biopsy procedures with up to 115 subjects at up to 10 centers.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Subject willing and able to comply with study procedures and provide written informed consent to participate in study.
3. Subject with a predominantly solid, peripheral lung lesion, 1 cm to 5 cm in diameter measured along its longest cross sectional diameter on axial CT imaging (obtained within 4 weeks per standard of practice) with the intention to undergo a clinically indicated bronchoscopic evaluation under routine clinical care. If the lesion is partially solid (i.e. there is a ground glass component) then the solid portion must make up at least 80% of the lesion.

   a. "Peripheral" lesion in this study will be pragmatically defined as any lesion in the lung parenchyma that the clinician feels cannot be accessed successfully using the convex probe endobronchial ultrasound bronchoscope.
4. Subject for whom the decision to pursue biopsy has been made by the treating physician and agreed upon by the subject.

Exclusion Criteria:

1. Subjects with pure ground glass opacity or a subsolid target lesion, and/or a ground glass opacity for which less than 80% of the lesion is solid identified by Chest CT.
2. Subjects who have medical contraindication to undergo conventional flexible or robotic bronchoscopy and standard of care Radial EBUS-guided cytological assessment evaluations, as determined by the investigator.
3. Subjects with known coagulopathy.
4. Subjects who are pregnant or nursing mothers.
5. Subjects who are currently enrolled in another investigational study that would directly interfere with the current study, without prior written approval from the sponsor.
6. Use of intraprocedural Cone Beam CT, Fixed CT or Augmented fluoroscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients where the needle is visualized by the iNOD system inside the lesion | Procedure
  Successful "Tool in lesion", defined as visualization of the tracheobronchial biopsy needle (TBNA) inside the targeted lesion within the ultrasound field of view.
Adverse Events | Procedure
  Proportion of subjects with Adverse Events related to the iNod device and/or study procedure, as well as Adverse Events related to any subsequent crossover procedures.

OTHER OUTCOMES:
Biopsy Yield | Procedure
  Diagnostic biopsy yield, defined as ability for histopathologist to report a specific benign or malignant diagnosis, stratified by concentric and eccentric lesion location.
Diagnostic Accuracy | 12 months post procedure
  Diagnostic accuracy at 12 months.
Device Rotation | Procedure
  Ability to reposition the needle into a different location within targeted lesions, if desired.
Crossover Rate | Procedure
  Crossover rate to radial EBUS or any alternative standard of care procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Chen, MD, Principal Investigator — Barnes-Jewish Hospital

IPD SHARING:
Plan to Share IPD: No